CLINICAL TRIAL: NCT01924520
Title: Phase I Study of FK949E - Phase I Oral Multiple-dose Study in Patients With Major Depressive Disorder
Brief Title: Oral Multiple-dose Study in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 6949-CL-0009
Record Dates: First submitted 2013-08-14; First posted 2013-08-16 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Major Depressive Disorder
Keywords: Antipsychotic; FK949E; Quetiapine
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (FK949E lower dose) (Experimental): Oral
  Interventions: Drug: FK949E
- Group 2 (FK949E middle dose) (Experimental): Oral
  Interventions: Drug: FK949E
- Group 3 (FK949E higher dose) (Experimental): Oral
  Interventions: Drug: FK949E

INTERVENTIONS:
Drug: FK949E — Oral
  Other Names: extended-release formulation of quetiapine

SUMMARY:
A study was to evaluate the safety and plasma concentration changes of quetiapine after repeated administration of FK949E (extended-release formulation of quetiapine) in patients with major depressive disorder (MDD).

DETAILED DESCRIPTION:
The objective of the study was to evaluate the safety and pharmacokinetics of multiple oral doses of FK949E (extended-release formulation of quetiapine) of three doses in patients with major depressive disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder by the M.I.N.I. according to the DSM-IV-TR
* Female patients of childbearing potential with a negative serum pregnancy test result and who were willing and able to use a reliable method of birth control during the study.
* Patients who could understand and comply with the requirements of the study, as judged by the investigator/sub-investigator.

Exclusion Criteria:

* A current or past history of a DSM-IV-TR Axis I disorder other than major depressive disorder within 6 months prior to provision of written informed consent.
* Diagnosis of a DSM-IV-TR Axis II disorder that was considered to have a major impact on the patient's current psychiatric status.
* A history of substance or alcohol abuse or dependence excluding caffeine and nicotine.
* Patients who were unable to abstain from drugs that induce or inhibit the drug-metabolizing enzyme CYP3A4 from 14 days prior to screening assessment and throughout the study period.
* Patients showing evidence or signs of renal or hepatic failure, serious heart disease, cerebrovascular disease, viral hepatitis B or C, or acquired immunodeficiency syndrome (AIDS) (carrier).
* Patients being treated for hypertension or patients with clinical finding that in the opinion of the investigator/sub-investigator could be negatively affected by the study or that would affect the study results (e.g., hypertension, unstable angina).
* Patients with concomitant hypotension or orthostatic hypotension (hypotension is defined as systolic blood pressure of less than 100 mmHg)
* Conditions that could affect absorption and metabolism of the study medication (e.g., malabsorption syndrome, liver disease)
* A current diagnosis of malignant tumor unless in remission for at least 5 years (except basal or squamous cell skin carcinoma).
* A history of transient ischemic attack (TIA).
* A history of seizure disorder, except for febrile convulsions
* Application of electroconvulsive therapy within 90 days prior to the start of study drug administration
* Use of a depot antipsychotic injection and inability to be off the drug for a period of twice the dosing interval prior to screening assessment and throughout the study period
* A score of ≥ 3 on the HAM-D17 Item (suicide) or a suicide attempt within the past 6 months. Patients judged to be at serious suicidal or homicidal risk in the opinion of the investigator/sub-investigator.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of unchanged quetiapine | for 24 hours after dosing
AUC24h (area under the curve for 24hr) of unchanged quetiapine | for 24 hours after dosing

SECONDARY OUTCOMES:
trough value of plasma concentration of unchanged quetiapine | for 24 hours after dosing
t1/2 of plasma concentration of unchanged quetiapine | for 24 hours after dosing
Maximum plasma concentration (Cmax) of quetiapine metabolites | for 24 hours after dosing
AUC (area under the curve) of quetiapine metabolites | for 24 hours after dosing
trough value of plasma concentration of quetiapine metabolites | for 24 hours after dosing
tmax of plasma concentration of quetiapine metabolites | for 24 hours after dosing
t1/2 of plasma concentration of quetiapine metabolites | for 24 hours after dosing
Safety assessed by the incidence of adverse events, clinical tab tests, vital signs, 12-lead ECGs and physical exam | Up to Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (2):
- Japan (2):
  - Kansai
  - Kantou

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=179